CLINICAL TRIAL: NCT06953635
Title: Quadratus Lumborum Blocks for Pain Control Following Open Ventral Hernia Repair: A Double Blinded Randomized Control Trial
Brief Title: Quadratus Lumborum Versus Placebo in Open Ventral Hernia Repair
Acronym: VHR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5342
Record Dates: First submitted 2025-01-24; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-03

CONDITIONS: Hernia, Ventral; Pain Management
Keywords: Regional Anesthesia; Postoperative Pain; Ventral Hernia Repair
MeSH Terms: conditions — Hernia, Ventral; Agnosia; Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: Study Design This is a prospective, double-blinded, randomized, placebo-controlled clinical trial comparing QL blocks to placebo for pain control for patients undergoing open VHR.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): The control (placebo comparator) group will undergo the same QL block procedure as the intervention arm, except saline (placebo) will be injected.
  Interventions: Procedure: Placebo
- Quadratus Lumborum Block (Experimental): The Quadratus Lumborum block will be randomly administered to half of the study patients.
  Interventions: Procedure: Quadratus Lumborum (QL) Block

INTERVENTIONS:
Procedure: Quadratus Lumborum (QL) Block — The intervention arm will receive bilateral quadratus lumborum blocks in the preoperative holding area prior to surgery. The syringe will contain a total of 60 mL of 0.25% Ropivacaine with 4 mg of Decadron. The anesthesiology pain team provider will administer 30 mL on the left side and 30 mL on the right side of the abdominal wall. The patient will receive one injection site per flank. During the procedure, the patient is placed in the left and then right lateral decubitus position and the ultrasound probe is placed above the iliac crest at the mid axillary line. The pain team provider will move the probe posteriorly to identify the "shamrock sign." Under ultrasound guidance, a needle is inserted in an in- plane approach through the quadratus lumborum (QL) muscle until reaching the middle of the thoracolumbar fascia layer between QL and psoas muscle. After negative aspiration for blood, injection will allow the spread of local anesthetic between the QL and psoas muscle on each side.
  Arms: Quadratus Lumborum Block
Procedure: Placebo — The placebo control group will receive the same quadratus lumborum (QL) block procedure as the intervention group, with the only difference being the injection of 60 mL of saline instead of local anesthetic. The anesthesiology team will administer 30 mL on each side of the abdominal wall, with one injection site per flank. The patient will be positioned in the left and right lateral decubitus positions, and the ultrasound probe will be placed above the iliac crest at the mid-axillary line to identify the "shamrock sign." The needle will be inserted through the QL muscle to the thoracolumbar fascia layer, between the QL and psoas muscle. After negative aspiration for blood, saline will be injected, allowing spread between the QL and psoas muscle on each side.
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether using a QL block is better than placebo (a look-alike substance that contains no drug) in lowering the amount of opioids you need for pain relief in the first 24 hours and if it improves your recovery following a ventral hernia repair.

Participants will be asked to complete a questionnaire before surgery and again at their 30-day follow up. You will also be asked to complete a pain diary 24 hours after surgery and attend a follow-up visit approximately 30 days after surgery.

The following information will be collected from you or your medical record:

1. Pain medications given to you during surgery.
2. Pain medications prescribed to you after surgery, including medication name, dose, units, and frequency.
3. Pain levels during the first 24 hours after surgery.
4. Your total hospital length of stay after surgery.
5. Any complications that you may have experienced after surgery.
6. Demographic information, medical history as well as details about your hernia repair surgery.

DETAILED DESCRIPTION:
Quadratus Lumborum (QL) blocks have provided analgesia for abdominal surgery. These blocks involve ultrasound-guided local anesthetic injection deep into the anterior fascia of the quadratus lumborum into the thoracolumbar fascia, resulting in widespread abdominal and pelvic pain control. QL blocks extend that coverage from T4 to L1 in the paravertebral space. At this local institution, QL blocks have demonstrated the ability to provide complete sensory analgesia for most patients from T9-L1 up to an estimated 17 hours after surgery. Therefore the goal of this study is to evaluate the effectiveness of QL block in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Able to read and understand study procedures
3. Willing to participate and sign an informed consent form
4. Open approaches to ventral hernia repair
5. Clean (CDC Class I), clean-contaminated (CDC Class II)
6. Elective surgery
7. Mesh placed in the retromuscular position

Exclusion Criteria:

1. Dirty-Infected cases (CDC Class IV): Old traumatic wounds with retained devitalized tissue and those that involve existing clinical infection or perforated viscera
2. Patient has a contraindication to receiving the drug and/or procedure: allergy/sensitivity to the drug, coagulopathy, abdominal wall infection at the drug administration site, systemic infection, anatomical distortion, neuropathy
3. Emergent procedure
4. Mesh not placed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-01-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Post-operative Opioid Utilization | From the time of treatment until 24 hours after surgery
  Quantity of Post-Operative Opioid Consumption as Measured by Morphine Milliequivalents for 24 Hours After Surgery

SECONDARY OUTCOMES:
Numerical rating Pain Score | From the time of treatment through hospitalization completion, an average of 4 days.
  Patient-reported pain will be recorded by the nursing staff at a minimum once per day, every day from the time of surgery until the patient is discharged from the hospital, an average of 4 days.
  Patient-reported pain will be scored on the validated Numeric Rating Scale (NRS), where patients are asked to choose a number between 0 and 10 that best describes their level of pain with "0" meaning "no pain" (better outcome) and "10" meaning "worst pain imaginable" (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Kaela E Blake, MD, Principal Investigator — The University of Tennessee Graduate School of Medicine
Locations (1):
- The University of Tennessee Medical Center, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roy A, Bhoi D, Chhabra A, Mohan VK, Darlong V, Prasad G. Quadratus lumborum block vs. transversus abdominis plane block in laparoscopic trans-abdominal pre-peritoneal repair of inguinal hernia in adults: A randomised controlled trial. Indian J Anaesth. 2023 Feb;67(2):207-215. doi: 10.4103/ija.ija_304_22. Epub 2023 Feb 16. PMID 37091451
- [Result] Liu X, Song T, Chen X, Zhang J, Shan C, Chang L, Xu H. Quadratus lumborum block versus transversus abdominis plane block for postoperative analgesia in patients undergoing abdominal surgeries: a systematic review and meta-analysis of randomized controlled trials. BMC Anesthesiol. 2020 Mar 2;20(1):53. doi: 10.1186/s12871-020-00967-2. PMID 32122319
- [Result] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Result] Fiore JF Jr, El-Kefraoui C, Chay MA, Nguyen-Powanda P, Do U, Olleik G, Rajabiyazdi F, Kouyoumdjian A, Derksen A, Landry T, Amar-Zifkin A, Bergeron A, Ramanakumar AV, Martel M, Lee L, Baldini G, Feldman LS. Opioid versus opioid-free analgesia after surgical discharge: a systematic review and meta-analysis of randomised trials. Lancet. 2022 Jun 18;399(10343):2280-2293. doi: 10.1016/S0140-6736(22)00582-7. PMID 35717988
- [Result] Schlosser KA, Renshaw SM, Tamer RM, Strassels SA, Poulose BK. Ventral hernia repair: an increasing burden affecting abdominal core health. Hernia. 2023 Apr;27(2):415-421. doi: 10.1007/s10029-022-02707-6. Epub 2022 Dec 26. PMID 36571666

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT06953635/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT06953635/ICF_001.pdf